CLINICAL TRIAL: NCT07394504
Title: Effects of Turning Based Dual Task Training on Balance and Mild Cognitive Impairment in Diabetic Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/29
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Neuropathy; Balance; Cognitive Dysfunction; Cognitive Decline
Keywords: Dual-task training; Dual-task Exercises
MeSH Terms: conditions — Diabetic Neuropathies; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Turning Based Dual-Task Training (Experimental): Group A receives Turning Based Dual-Task Training:
  The intervention will be conducted over a total duration of 8 weeks with total of 24 sessions 3 days per week lasting for 30 to 40 minutes. Warm up, Conventional balance training and cool down.
  Interventions: Procedure: Turning Based Dual Task Training
- Dual-Task Training (Experimental): Group B receives Dual-Task Training:
  The intervention will be conducted over a total duration of 8 weeks with total of 24 sessions 3 days per week lasting for 30 to 40 minutes. Warm up, Conventional balance training and cool down.
  Interventions: Procedure: Dual-Task Training

INTERVENTIONS:
Procedure: Turning Based Dual Task Training — Intervention will be of 8 weeks , 24 sessions, three per week, lasting 30-40 minutes. Warm-up exercises followed by cool down.
  Conventional balance training consisting sitting eyes open/closed, dynamic weight shifting, Static/tandem Standing.
  Turning protocol will be in three progressive phases. Phase 1 will include turning around cone, obstacles, during walking and 8 figure walk with cognitive dual task( name animals, shapes etc). Phase 2 exercises are 360 turn, sudden turn, stepping with turn, 8 figure turn and obstacle turn with more cognitive load. Phase 3 exercises are all exercises above in tandem walk with reaching activites and more cognitive load.
  Arms: Turning Based Dual-Task Training
Procedure: Dual-Task Training — Intervention will be of 8 weeks , 24 sessions, three per week, lasting 30-40 minutes. Warm-up exercises followed by cool down.
  Conventional balance training consisting sitting eyes open/closed, dynamic weight shifting, Static/tandem Standing.
  This protocol will be in three progressive phases. Phase 1 will include sit to stand, dynamic weight shifting (standing), stepping, walking in multi direction with cognitive task like name countries, sentence completion etc. Phase 2 will include additional step over low obstacle in walking along the above exercises with more repetitions and increased cognitive load.
  Phase 3 will include tandem walk, step over high obstacle, ball throw/catch, multi direction walk in tandem with more increased cognitive load respectively.
  Arms: Dual-Task Training

SUMMARY:
Diabetic Peripheral Neuropathy (DPN) is a common complication of diabetes, characterized by impaired sensory and motor function, often leading to balance dysfunction and an increased risk of falls. Additionally, individuals with DPN are at heightened risk for mild cognitive impairment (MCI), which further compromises functional independence. This study aims to determine the effects of turning-based dual-task training compared to conventional dual-task training on balance, cognitive function, and fall risk in individuals with DPN. Pre- and post-intervention assessments will be conducted using the Berg Balance Scale (BBS), Montreal Cognitive Assessment (MoCA), and Timed Up and Go Test (TUGT) to evaluate balance, cognition, and fall risk respectively.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a chronic metabolic disorder characterized by hyperglycemia resulting from defects in insulin secretion, insulin action or both. As a major global health concern, its prevalence has been steadily increasing. According to the recent searches, 26.7% of adults in Pakistan are affected by diabetes. Implicated poor glycemic control, duration of diabetes, hyperlipidemia (particularly hypertriglyceridemia), elevated albumin excretion rates and obesity as risk factors for the development of DPN. This study aims to explore the effectiveness of these interventions in this specific population and to tell a treatment that will target both balance and cognition that will be used for DPN patients to improve the symptoms.

A randomized controlled trial will be conducted over one year. 44 participants will be selected through non- probability purposive sampling and randomly divided into two groups. The intervention will last eight weeks, comprising 24 treatment sessions. Assessments will be conducted at baseline and at the end of eight week. Treatment for Group A will include warm up, conventional balance training, turning based dual task training followed by cool down. Group B will include warm up, conventional balance training, dual task training followed by cool down.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus ≥ 5 years
* Diagnosed with Diabetic Peripheral Neuropathy
* Age 50 and above
* Berg Balance Scale (BBS 21-40) score
* Mild Cognitive Impairments (MoCA 18-25)
* Able to stand and walk with or without assistive devices

Exclusion Criteria:

* Severe neuropathic foot ulcers or Charcot joints.
* History of major musculoskeletal injuries affecting ambulation (Fractures of lower limb), Severe Osteoarthritis.
* Uncontrolled Diabetes.
* Neurological disorders unrelated to DPN (brain tumors, stroke, epilepsy, Alzheimer's, GBS and Parkinson's disease).
* Significant visual, auditory impairment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Balance | 8 weeks
  Balance is assessed by Berg Balance Scale. Interpretations: mild=41-56,moderate=21-40,severe=0-20
Cognition | 8 weeks
  MoCA will be used for mild cognitive impairment. Interpretations: Mild= 18-25, Moderate=10-17, Severe=0-9
Fall Risk | 8 weeks
  Timed up and go test will be used for Fall Risk. Interpretations: Low Risk: <10 seconds, Moderate Risk: 10-19 seconds, High Risk: ≥ 14-20 seconds, Severe Risk: > 30 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan